CLINICAL TRIAL: NCT05907421
Title: Altered Neural Activation Patterns During Emotion Regulation in Adolescents With Nonsuicidal Self-Injury Under Naturalistic Immersive Emotional Engagement
Brief Title: Emotion Regulation Dysfunctions in NSSI Adolescents in Naturalistic Contexts
Status: Recruiting | Type: Observational
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Other Study IDs: BAM_lab_NSSI_01
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nonsuicidal Self Injury; Emotion Regulation
MeSH Terms: conditions — Self-Injurious Behavior; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSSI
  Interventions: Behavioral: Acceptance mindset
- HC
  Interventions: Behavioral: Acceptance mindset

INTERVENTIONS:
Behavioral: Acceptance mindset — Brief training of acceptance versus emotional reactivity as emotion regulation strategy.

SUMMARY:
Nonsuicidal self-injury (NSSI) is defined as direct, deliberate bodily harm without suicidal intention. Recent studies indicate that prevalence rates are increasing worldwide, in particular under adolescents, indicating a growing public health issue. An impaired ability to regulate negative emotion has been suggested to play a potential role in NSSI behavior. Some recent interventions aim at improving dysfunctional emotion regulation via 'acceptance'. Acceptance represents an objective, nonreactive, nonjudgmental, and calming emotion regulation strategy, partly based on the philosophy of dialectical behavior therapy (DBT) that has been widely used in the clinical treatment of NSSI behaviors. The aim of the present functional magnetic resonance imaging (fMRI) study is to examine whether adolescents with NSSI can implement the acceptance strategy in naturalistic emotional contexts (immersive video clips) and whether they differ from healthy controls in terms of behavioral and neural effects. To this end, the investigators recruit one group of NSSI adolescents (n=40) and one healthy control group (n=40), to compare the subjective emotional experience as well as underlying neural activity as measured by blood oxygenation level-dependent (BOLD) fMRI. The investigators hypothesize that compared to HC, NSSI adolescents will experience stronger negative emotions and show dysregulated neural recruitment of brain systems engaged in emotional reactivity and regulations (e.g. limbic regions, default mode network, and frontal regions).

ELIGIBILITY:
Inclusion Criteria:

* 15-18 years
* right-handed
* normal or corrected normal visual acuity
* meet the proposed DSM-5 frequency criteria (e.g., ≥5 days of NSSI behaviors in the past year)

Exclusion Criteria:

* diagnosis of borderline personality disorder, major depressive disorder, other psychiatric disorders, etc.
* high suicidal risk
* recent use of medications that can affect neural activity
* have received or are receiving Dialectical Behavior Therapy (DBT) other treatment for emotional problems within the past 6 months
* have a contraindication to MRI scanning (e.g., metal implants, claustrophobia or other conditions that make them inappropriate for MRI scanning)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Treatment-seeking NSSI individuals will be recruited from local hospitals and HC from the community.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Negative subjective emotional experience as indexed by self-report | About 30 minutes
  Subjects will rate their negative affect on a scale ranging from 1-9 in response to neutral and negative emotional stimuli during normal experience or acceptance. Alterations in the patients will be determined by using ANOVA models with the group (NSSI vs. HC) as a between-subject factor and emotion regulation condition as a within-subject factor.
Neural activity as indexed by BOLD fMRI | About 30 minutes
  Brain activity will be monitored by task-based fMRI. Alterations in the patients will be determined by the experimental groups (NSSI vs. HC) with respect to the emotion regulation conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial Center for Mental Health, Sichuan Provincial People's Hospital, University of Electronic Science and Technology of China, Chengdu, Sichuan, China